CLINICAL TRIAL: NCT05587062
Title: A Phase III, Multicenter, Randomized, Two-armed, Double-blind, Parallel, Active-controlled, Non-inferiority Clinical Trial to Compare Efficacy and Safety of Aflibercept (CinnaGen Co, Iran) to the Reference Aflibercept Product (Eylea®, Regeneron, USA) in Patients With Neovascular Age-related Macular Degeneration.
Brief Title: Efficacy and Safety of Aflibercept in Patients With Neovascular Age-related Macular Degeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN.AFL.RK.PH3.2018
Record Dates: First submitted 2022-09-18; First posted 2022-10-19 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Age-Related Macular Degeneration; Neovascular Age-related Macular Degeneration
Keywords: AMD; nAMD; Recombinant Fusion Protein; anti-VEGF; Aflibercept
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aflibercept (CinnaGen Co, Iran) (Experimental): Aflibercept (CinnaGen Co, Iran) 2 mg (0.05 mL) by intravitreal injection every 4 weeks for the first 3 injections, followed by 2 mg every 8 weeks until week 48 of study
  Interventions: Biological: Aflibercept (CinnaGen Co, Iran)
- Aflibercept (Regeneron, USA) (Active Comparator): Aflibercept (Regeneron, USA) 2 mg (0.05 mL) by intravitreal injection every 4 weeks for the first 3 injections, followed by 2 mg every 8 weeks until week 48 of study
  Interventions: Biological: Aflibercept (Regeneron, USA)

INTERVENTIONS:
Biological: Aflibercept (CinnaGen Co, Iran) — Aflibercept (CinnaGen Co, Iran) by intravitreal injection
  Arms: Aflibercept (CinnaGen Co, Iran)
Biological: Aflibercept (Regeneron, USA) — Aflibercept (Regeneron, USA) by intravitreal injection
  Other Names: Eylea®
  Arms: Aflibercept (Regeneron, USA)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Aflibercept (produced by CinnaGen Co, Iran) compared with Eylea® (Regeneron, USA) in subjects with Neovascular Age-related Macular Degeneration (nAMD).

All the participants will receive one of the following regimens:

Aflibercept (CinnaGen Co, Iran) or Eylea® (Regeneron, USA), 2 mg (vial 0.05 ml) by intravitreal injection every 4 weeks for the first 3 injections, followed by 2 mg every 8 weeks until week 48 of study.

The primary objective of this study is to verify the non-inferiority of Aflibercept (CinnaGen Co, Iran) versus Eylea® (Regeneron, USA) in achieving maintaining vision (losing<15 letter on ETDRS chart) at week 52 in comparison to week 0 in participants with Neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 55-80 years at the time of signing the informed consent form.
2. Primary active CNV subfoveal lesion secondary to AMD, with definite diagnosis of AMD, according to the physician's decision, based on the results of ocular examination, or OCT, based on the following diagnostic Criteria:

   • Evaluating the presence of Submacular hemorrhage in fundus examination with the presence of any of those items mentioned in OCT including: subretinal fluid, subretinal hyper reflective material, intraretinal fluid or pigment epithelial detachment.

   Or

   • Diagnosis of the following, based on the OCT evaluations:
   * Presence of pigment epithelial detachment with intra-retinal fluid and subretinal fluid
   * Presence of pigment epithelial detachment with intra-retinal fluid and subretinal hyper reflective material

   The presence of new vessels should be confirmed with one of the additional imaging modalities (FA or ICG or OCTA).

   In cases with any suspicious for the diagnosis of AMD, other confirmatory modalities should be used.
3. The ETDRS-best-corrected visual acuity index with the score of 20/40 to 20/320 (or BCVA letter score of 73 to 25 in the study eye), which is determined by a specific trained person, within the standard distance, in each study center.
4. Willing, committed, and able to return for clinic visits and complete all study-related procedures.
5. Patients with the ability to read, (or, if unable to read due to visual impairment, be read by a family member or person administering the informed consent form) understand and willing to sign the informed consent form for participation in the study.

Exclusion Criteria:

1. Any prior ocular or systemic anti-VEGF therapy, during the past three months, Photodynamic Therapy (PDT) or surgery for neovascular AMD.
2. The need for receiving ocular anti-VEGF simultaneously in both eyes in the loading phase for the treatment of neovascular AMD (in fact, if the patient, in addition to the study eye, also needs to receive the drug for the opposite eye)
3. Scar, fibrosis, or extensive subretinal hemorrhage of more than 50% of the total lesion area in the study eye, according to the physician's opinion based on clinical presentation or according to fundus photography.
4. The presence of scar, fibrosis, or atrophy in the central part of the fovea in the study eye.
5. The presence of retinal pigment epithelial tears or rips involving the macular part of the study eye at the time of entering the study.
6. The history of any vitreous hemorrhage within four weeks prior to the first visit of the study in the study eye.
7. Presence of other causes of CNV, including pathologic myopia (spherical equivalent of -8 diopters or more negative, or axial length of 25 mm or more), ocular histoplasmosis syndrome, angioid streaks, choroidal rupture, or multifocal choroiditis in the study eye.
8. Clinical or paraclinical diagnosis of PCV by the physician at baseline
9. The history or clinical evidence of diabetic retinopathy, diabetic macular edema, or any other vascular disease affecting the retina, other than AMD in either eyes.
10. Prior vitrectomy in the study eye.
11. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
12. Any history of a macular hole of stage two or above in the study eye.
13. Any intraocular or periocular surgery within three months of the screening visit on the study eye except lid surgery, which may not have taken place within one month of screening visit, as long as it's unlikely to interfere with the injection during the study.
14. Prior trabeculectomy or any other filtration surgery in the study eye.
15. Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication) in the study eye.
16. Active intraocular inflammation in either eye.
17. Active ocular or periocular infection in either eye
18. Any ocular or periocular infection within the last two weeks prior to screening visit in either eye.
19. Any history of uveitis in either eye.
20. Presence or history of scleromalacia in either eye.
21. Aphakia or pseudophakia with the absence of posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] posterior capsulotomy) in the study eye.
22. Previous therapeutic radiation in the region of the study eye.
23. History of corneal transplant or corneal dystrophy in the study eye.
24. Any significant media opacities, including cataract, in the study eye that might interfere with visual acuity, assessment of drug safety, or fundus photography.
25. Patients with amblyopia.
26. Patients with blindness in the opposite eye (if for any reason, the patient's vision in the opposite eye is limited to understanding the light and movement of the hands, the patient should not enter the study, but if the best-corrected visual acuity index is 20/400 or more, it is not a problem).
27. Any concurrent intraocular condition in the study eye that, in the opinion of the investigator, could require either medical or surgical intervention during the study period.
28. Any concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the patient beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of efficacy or safety.
29. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the patient at high risk for treatment complications.
30. Participation as a patient in any clinical study within the 12 weeks prior to the screening visit.
31. The use of long-acting steroids, either systemically or intraocularly, in the six months prior to screening visit.
32. Any history of allergy to povidone iodine.
33. Females who are pregnant, breastfeeding, planning to become pregnant during the study period, unwilling to practice adequate contraception throughout the study and for at least 60 days following the last dose of study medication.
34. History of stroke, myocardial infarction or uncontrolled hypertension (blood pressure >160/100 despite receiving medical treatment) for less than three months from the date of the Screening visit.
35. Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients achieving maintaining vision at week 52 | At week 52
  Achieving maintaining vision confirmed by losing<15 letter on ETDRS chart

SECONDARY OUTCOMES:
Mean changes in the Best-Corrected Visual Acuity Index from week 0 to week 52 | Baseline and at week 52
  Changes in Best-Corrected Visual Acuity Index measured with ETDRS chart
The percentage of patients who have increase of ≥15 score in ETDRS at week 52 compared to week 0 | Baseline and at week 52
  Increase of ≥15 score in ETDRS chart demonstrates improvement in visual function
The mean change in National Eye Institute Visual Function Questionnaire (NEI VFQ-25) at week 52 compared to week 0 | Baseline and at week 52
  The NEI VFQ-25 (National Eye Institute Visual Functioning Questionnaire) is a self-reported vision-targeted health status which has importance value in chronic eye diseases. Total score range is from 0 to 100. In this scale, score of 0 demonstrates the worst outcome and 100 means the best outcome. The NEI VFQ -25 has a collection of subscales which are all scored from 0-100. The overall score is average of all subscale in order to give each sub-scale equal weight.
Mean changes in central retinal thickness at week 52 compared to the screening visit | Baseline and at week 52
  Retinal thickness is measured by Optical Coherence Tomography (OCT) which shows disease activity in Neovascular Age-related Macular Degeneration
The percentage of patients without intra-retinal fluid and subretinal fluid at week 52 | Baseline and at week 52
  Intra-retinal fluid and subretinal fluid measured with Optical Coherence Tomography (OCT)
Number of participants with Adverse Events (AEs) | Baseline up to Week 52
  Systemic and ophthalmic Adverse Events (AEs) and Adverse Drug Reactions (ADR) at baseline, all the visits to the end of week 52, evaluation of vital sign including blood pressure and physical examination findings at baseline and at week 52, clinical laboratory testing including liver and kidney functions, complete blood count, and clinical bio-chemistries and immunogenicity assessment at baseline, week 24 and week 52

CONTACTS AND LOCATIONS:
Locations (1):
- Farabi Hospital, Tehran, Iran